CLINICAL TRIAL: NCT00161304
Title: Effects of Testosterone Administration on Tissues of Men With A.D.A.M. (Androgen Deficiency of Aging Men)
Brief Title: Study to Determine the Effects of Testosterone Replacement Therapy in Aging Men With Androgen Deficiency
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Leonard S. Marks, M.D. (Other)
Collaborators: Solvay Pharmaceuticals (Industry); Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Leonard S. Marks, M.D., Principal Investigator, Urological Sciences Research Foundation
Organization: Urological Sciences Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T-001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Men With Low Testosterone Levels
MeSH Terms: interventions — testosterone enanthate; Testosterone

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Testosterone Enanthate (Active Comparator): Testosterone
  Interventions: Drug: Testosterone Enanthate
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Testosterone Enanthate — Testosterone Enanthate
  Other Names: testosterone
  Arms: Testosterone Enanthate
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
The T-001 study is a placebo-controlled investigation of the effects of injectable testosterone replacement therapy on prostate tissues of aging men with low testosterone levels.

DETAILED DESCRIPTION:
The T-001 study is a placebo-controlled investigation of the effects of injectable testosterone replacement therapy on prostate tissues of aging men with low testosterone levels. The primary objectives of the study are to measure the changes in tissue hormones and other biomarkers in the prostate tissue specimens.

ELIGIBILITY:
The screening evaluation consisted of:

1. medical history, which included the androgen deficiency of the aging male questionnaire
2. physical examination
3. multiphasic serum panel
4. measurement of total serum testosterone and PSA levels

Exclusion criteria included:

1. use in the past 6 months of any drug potentially affecting the pituitary-gonadal axis
2. serum PSA level greater than 10.0 ng/mL
3. refusal or inability to undergo prostate biopsies
4. presence of prostate cancer on initial biopsy results.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-04 (Actual); Primary Completion 2004-08 (Actual); Study Completion 2004-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard S Marks, M.D., Principal Investigator — Urological Sciences Research Foundation
Locations (1):
- Urological Sciences Research Foundation, Culver City, California, United States

REFERENCES:
- [Derived] Marks LS, Mazer NA, Mostaghel E, Hess DL, Dorey FJ, Epstein JI, Veltri RW, Makarov DV, Partin AW, Bostwick DG, Macairan ML, Nelson PS. Effect of testosterone replacement therapy on prostate tissue in men with late-onset hypogonadism: a randomized controlled trial. JAMA. 2006 Nov 15;296(19):2351-61. doi: 10.1001/jama.296.19.2351. PMID 17105798
- See also: Urological Sciences Research Foundation — http://www.usrf.org